CLINICAL TRIAL: NCT01672879
Title: A Phase 2b, Dose-Ranging, Randomized, Double-Blind, Placebo-Controlled Trial Evaluating the Safety and Efficacy of GS-6624, a Monoclonal Antibody Against Lysyl Oxidase-Like 2 (LOXL2), in Subjects With Compensated Cirrhosis Secondary to Non-Alcoholic Steatohepatitis (NASH)
Brief Title: Simtuzumab (SIM, GS-6624) in the Treatment of Cirrhosis Due to NASH
Acronym: NASH
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GS-US-321-0106; 2012-002489-11 (EudraCT Number)
Record Dates: First submitted 2012-08-22; First posted 2012-08-27 (Estimated); Results first posted 2019-03-27 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Liver Fibrosis Due to NASH
Keywords: NASH; cirrhosis; Compensated Liver disease; Monoclonal antibody; LOXL2; Simtuzumab; Nonalcoholic Steatohepatitis; Hepatic venous pressure gradient; HVPG; NAFLD; MRE; Liver biopsy; Liver fibrosis; Ishak
MeSH Terms: conditions — Fibrosis; Non-alcoholic Fatty Liver Disease; Liver Cirrhosis | interventions — simtuzumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- SIM 200 mg (Experimental): During the Randomized Double-Blind Phase, participants will receive SIM 200 mg via intravenous infusion every 2 weeks for up to 240 weeks. During the optional Open-Label Phase, participants will receive SIM 700 mg via intravenous infusion every 2 weeks for up to an additional 240 weeks.
  Interventions: Biological: SIM
- SIM 700 mg (Experimental): During the Randomized Double-Blind Phase, participants will receive SIM 700 mg via intravenous infusion every 2 weeks for up to 240 weeks. During the optional Open-Label Phase, participants will receive SIM 700 mg via intravenous infusion every 2 weeks for up to an additional 240 weeks.
  Interventions: Biological: SIM
- Placebo (Placebo Comparator): During the Randomized Double-Blind Phase, participants will receive placebo to match SIM administered via intravenous infusion every 2 weeks for up to 240 weeks. During the optional Open-Label Phase, participants will receive SIM 700 mg administered via intravenous infusion every 2 weeks for up to an additional 240 weeks.
  Interventions: Biological: Placebo; Biological: SIM

INTERVENTIONS:
Biological: Placebo — Placebo to match SIM intravenous infusion over 30 minutes every 2 weeks
  Arms: Placebo
Biological: SIM — Intravenous infusion over 30 minutes every 2 weeks
  Other Names: GS-6624

SUMMARY:
The primary objective of this study is to evaluate the safety and efficacy of SIM (formerly referred to as GS-6624) in adults with compensated cirrhosis due to Non-Alcoholic Steatohepatitis (NASH). It will consist of 2 phases:

* Randomized Double-Blind Phase
* Open-Label Phase (optional)

ELIGIBILITY:
Key Inclusion Criteria:

* Adults with cirrhosis of the liver defined as an Ishak fibrosis stage ≥ 5
* Liver biopsy consistent with NASH or cryptogenic cirrhosis
* Exclusion of other causes of liver disease including viral hepatitis and alcoholic liver disease
* The liver biopsy sample must be determined to be adequate for evaluation by the Central pathologist
* Must have aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 10 x the upper limit of the normal range (ULN)
* Must have serum creatinine < 2.0 mg/dL
* A negative serum pregnancy test is required for female subjects of childbearing potential
* All sexually active female subjects of childbearing potential must agree to use a protocol recommended method of contraception during heterosexual intercourse throughout the study and for 90 days following the last dose of study medication
* Lactating females must agree to discontinue nursing before starting study treatment
* Male subjects, if not vasectomized, are required to use barrier contraception (condom plus spermicide) during heterosexual intercourse from the screening through the study completion and for 90 days following the last dose of study drug

Key Exclusion Criteria:

* Pregnant or breast feeding
* Any history of hepatic decompensation including ascites, hepatic encephalopathy or variceal bleeding
* Weight reduction surgery in the past 5 year
* Child-Pugh-Turcotte (CPT) score >7; Model for End-Stage Liver Disease (MELD) score > 12 and Body Mass Index (BMI) <18kg/m2
* Positive for hepatitis C virus (HCV) RNA
* Positive for HBsAg
* Alcohol consumption greater than 21oz/week for males or 14oz/week for females
* Positive urine screen for amphetamines, cocaine or opiates (i.e. heroin, morphine) at screening. Subjects on stable methadone or buprenorphine maintenance treatment for at least 6 months prior to screening may be included in the study. Subjects with a positive urine drug screen due to prescription opioid-based medication are eligible if the prescription and diagnosis are reviewed and approved by the investigator
* Clinically significant cardiac disease
* History of malignancy, other than non-melanomatous skin cancer, within 5 years prior to screening
* Major surgical procedure within 30 days prior to screening or the presence of an open wound
* Known hypersensitivity to the investigation product or any of its formulation excipients
* History of bleeding diathesis within 6 months of screening
* Unavailable for follow-up assessment or concern for subject's compliance with the protocol procedures;
* Participation in an investigational trial of a drug or device within 30 days prior to screening
* History of solid-organ transplant; poor venous access or requirement for permanent or semi-permanent central vein catheter such as portacath

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 259 (Actual)
Dates: Start 2012-10-29 (Actual); Primary Completion 2016-09-26 (Actual); Study Completion 2017-01-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (59):
- United States (41):
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Southern California Liver Centers, Coronado, California
  - University of California, San Diego (UCSD), San Diego, California
  - University of California San Francisco (UCSF), San Francisco, California
  - University of Colorado, Denver, Aurora, Colorado
  - University of Miami, Miami, Florida
  - Tampa General Hospital, Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - Indiana University School of Medicine, Division of Gastroenterology/Hepatology, Indianapolis, Indiana
  - Iowa Digestive Disease Center, Clive, Iowa
  - University of Louisville, Louisville, Kentucky
  - Tulane University, New Orleans, Louisiana
  - Mercy Medical Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Lahey Clinic, Burlington, Massachusetts
  - University of Mississippi Medical Center, Jackson, Michigan
  - Minnnesota Gastroenterology, PA, Saint Paul, Minnesota
  - Saint Louis University Hospital, St Louis, Missouri
  - State University Of New York at Buffalo, Buffalo, New York
  - North Shore University Health System, Manhasset, New York
  - New York University, New York, New York
  - Columbia University Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - University of Pennsylvania Hospital, Philadelphia, Pennsylvania
  - University Gastroenterology, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Methodist University Hospital, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Clinical Research Institute, Arlington, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - St. Luke Episcopal Hospital, Houston, Texas
  - Alamo Clinical Research Associates, San Antonio, Texas
  - Intermountain Transplant Center, Murray, Utah
  - University of Virginia Health Center, Charlottesville, Virginia
  - Liver Institute of Virginia, Newport News, Virginia
  - Digestive and Liver Disease Specialists, Norfolk, Virginia
  - Bucheon St. Marys Hospital, Richmond, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - University of Washington, Seattle, Washington
- Canada (3):
  - University of Manitoba, Winnipeg, Manitoba
  - Dalhousie University, Halifax, Nova Scotia
  - Toronto Liver Centre, Toronto, Ontario
- France (4):
  - Hôpital de la Croix Rousse, Lyon
  - Hospital Saint-Antoine, Paris
  - CHU Pitié-Salpêtrière, Paris
  - Fonds de Recherche Honoraires, Strasbourg
- Germany (2):
  - Gastroenterologisch-Hepatologisches Zentrum Kiel, Kiel
  - Eugastro Gmbh, Leipzig
- Italy (3):
  - Istituto Clinico Humanitas, Rozzano, Milano
  - Azienda Ospedaliero-Universitaria Policlinico di Modena, Modena
  - Azienda Ospedaliera Città della Salute e della Scienza di Torino, Torino
- Fundacion De Investigacion, San Juan, Puerto Rico
- Spain (2):
  - Hospital Vall D´Hebron, Barcelona, Catalonia
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
- United Kingdom (3):
  - Royal Free Hospital, Pond Street, London
  - King's College Hospital NHS Trust, London
  - Nottingham University Hospitals Queen's Medical Centre, Nottingham

REFERENCES:
- [Result] Sanyal A, Harrison S, Ratziu V, Abdelmalek M, Diehl A, Caldwell S, et al. Changes in fibrosis, but not the NAFLD Activity Score (NAS), are associated with disease progression in patients with nonalcoholic steatohepatitis (NASH) and advanced fibrosis. J Hepatol 2017; 66 (1): S2.
- [Result] Sanyal A, Abdelmalek M, Diehl A, Caldwell S, Shiffman M, Ghalib R, et al. Efficacy and safety of simtuzumab for the treatment of nonalcoholic steatohepatitis with bridging fibrosis or cirrhosis: results of two phase 2b, dose-ranging, randomized, placebo-controlled trials. J Hepatol 2017; 66 (1): S54.
- [Result] Bosch J, Harrison S, Ratziu V, Shiffman M, Diehl A, Caldwell S, et al. Impact of modest weight reduction on liver histology, portal pressure, and clinical events in patients with compensated cirrhosis due to nonalcoholic steatohepatitis. J Hepatol 2017; 66 (1): S159-S160.
- [Result] Sanyal A, Goodman Z, Harrison S, Rockey DC, Diehl AM, Caldwell S, et al. Correlation between the hepatic venous pressure gradient and alpha-smooth muscle actin (SMA) expression in patients with compensated cirrhosis due to nonalcoholic steatohepatitis. J Hepatol 2016; 64 (2): S251.
- [Result] Shea PR, Sanyal A, Harrison S, Ratziu V, Loomba R, Caldwell S, et al. PNPLA3 variants confer an increased risk of advanced fibrosis due to non-alcoholic steatohepatitis. J Hepatol 2016; 64 (2): S493.
- [Result] Shea PR, Sanyal A, Rockey DC, Loomba R, Diehl AM, Kleinstein SE, et al. Genome-wide association study of clinically significant portal hypertension in patients with nonalcoholic steatohepatitis and advanced fibrosis. J Hepatol 2016; 64 (2): S280.
- [Result] Bosch J, Ratziu V, Rockey DC, Ghalib RH, Thuluvath PJ, Shiefke I, et al. Correlation between noninvasive markers of fibrosis and the hepatic venous pressure gradient (HVPG) in patients with compensated cirrhosis due to nonalcoholic steatohepatitis (NASH). Hepatol 2015; 62 (1): 578A.
- [Result] Goodman ZD, Alaparthi L, Monge F, Patel K, Loomba R, Caldwell SH, et al. Correlations between hepatic morphometric collagen content, histologic fibrosis staging, and serum markers in patients with advanced fibrosis due to nonalcoholic steatohepatitis (NASH). Hepatol 2015; 62 (1): 906A.
- [Result] Harrison SA, Goodman ZD, Ratziu V, Loomba R, Diehl AM, Lawitz E, et al. Serum lysyl oxidase-like-2 (sLOXL2) levels correlate with fibrosis stage in patients with nonalcoholic steatohepatitis (NASH). Hepatol 2015; 62 (1): 910A.
- [Result] Sanyal AJ, Goodman ZD, Abdelmalek MF, Harrison SA, Rockey DC, Diehl AM, et al. Clinical and histologic correlates of the hepatic venous pressure gradient (HVPG) in patients with compensated cirrhosis due to nonalcoholic steatohepatitis (NASH). Hepatol 2015; 62 (1): 577A.
- [Result] Ratziu V, Sanyal AJ, Loomba R, Caldwell SH, Ghalib RH, Torres DM, et al. Characterization of insulin resistance in patients with advanced fibrosis due to nonalcoholic steatohepatitis (NASH). Hepatol 2015; 62 (1): 1298A-1299A.
- [Derived] Loomba R, Huang DQ, Sanyal AJ, Anstee QM, Trauner M, Lawitz EJ, Ding D, Ma L, Jia C, Billin A, Huss RS, Chung C, Goodman Z, Wong VW, Okanoue T, Romero-Gomez M, Abdelmalek MF, Muir A, Afdhal N, Bosch J, Harrison S, Younossi ZM, Myers RP. Liver stiffness thresholds to predict disease progression and clinical outcomes in bridging fibrosis and cirrhosis. Gut. 2023 Mar;72(3):581-589. doi: 10.1136/gutjnl-2022-327777. Epub 2022 Sep 9. PMID 36750244
- [Derived] Younossi ZM, Anstee QM, Wai-Sun Wong V, Trauner M, Lawitz EJ, Harrison SA, Camargo M, Kersey K, Subramanian GM, Myers RP, Stepanova M. The Association of Histologic and Noninvasive Tests With Adverse Clinical and Patient-Reported Outcomes in Patients With Advanced Fibrosis Due to Nonalcoholic Steatohepatitis. Gastroenterology. 2021 Apr;160(5):1608-1619.e13. doi: 10.1053/j.gastro.2020.12.003. Epub 2020 Dec 8. PMID 33307033
- [Derived] Harrison SA, Abdelmalek MF, Caldwell S, Shiffman ML, Diehl AM, Ghalib R, Lawitz EJ, Rockey DC, Schall RA, Jia C, McColgan BJ, McHutchison JG, Subramanian GM, Myers RP, Younossi Z, Ratziu V, Muir AJ, Afdhal NH, Goodman Z, Bosch J, Sanyal AJ; GS-US-321-0105 and GS-US-321-0106 Investigators. Simtuzumab Is Ineffective for Patients With Bridging Fibrosis or Compensated Cirrhosis Caused by Nonalcoholic Steatohepatitis. Gastroenterology. 2018 Oct;155(4):1140-1153. doi: 10.1053/j.gastro.2018.07.006. Epub 2018 Jul 7. PMID 29990488

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Europe and North America. The first participant was screened on 29 October 2012. The last study visit occurred on 03 January 2017.
Pre-assignment Details: 453 participants were screened.
Groups:
- SIM 200 mg: Blinded Phase: Participants received simtuzumab (SIM) 200 mg administered via intravenous infusion every 2 weeks for up to 240 weeks.
  Open-Label Phase: Participants received SIM 700 mg administered via intravenous infusion every 2 weeks for up to an additional 240 weeks.
- SIM 700 mg: Blinded Phase: Participants received SIM 700 mg administered via intravenous infusion every 2 weeks for up to 240 weeks.
  Open-Label Phase: Participants received SIM 700 mg administered via intravenous infusion every 2 weeks for up to an additional 240 weeks.
- Placebo: Blinded Phase: Participants received placebo to match SIM administered via intravenous infusion every 2 weeks for up to 240 weeks.
  Open-Label Phase: Open-Label Phase: Participants received SIM 700 mg administered via intravenous infusion every 2 weeks for up to an additional 240 weeks.
Period: Blinded Phase (Up to 240 Weeks)
Arm/Group | SIM 200 mg | SIM 700 mg | Placebo
Started | 87 | 86 | 86
Completed | 0 | 0 | 0
Not Completed | 87 | 86 | 86
Not completed — Study Terminated by Sponsor | 43 | 55 | 61
Not completed — Withdrew Consent | 14 | 7 | 6
Not completed — Adverse Event | 5 | 2 | 7
Not completed — Lost to Follow-up | 4 | 3 | 1
Not completed — Investigator's Discretion | 5 | 0 | 2
Not completed — Death | 0 | 2 | 0
Not completed — Missing | 1 | 0 | 0
Not completed — Randomized but Never Treated | 0 | 0 | 1
Not completed — Met Protocol-Specified Reason(s) | 15 | 17 | 8
Period: Open-Label Phase (Up to 240 Weeks)
Arm/Group | SIM 200 mg | SIM 700 mg | Placebo
Started | 15 (Met protocol-specified reason(s) for study discontinuation during Blinded Phase & entered Open-Label) | 17 (Met protocol-specified reason(s) for study discontinuation during Blinded Phase & entered Open-Label) | 8 (Met protocol-specified reason(s) for study discontinuation during Blinded Phase & entered Open-Label)
Completed | 0 | 0 | 0
Not Completed | 15 | 17 | 8
Not completed — Study Terminated by Sponsor | 8 | 16 | 6
Not completed — Adverse Event | 5 | 1 | 1
Not completed — Investigator's Discretion | 1 | 0 | 1
Not completed — Progressive Disease | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all enrolled participants who were randomized and received at least one dose of study drug.
Groups:
- SIM 200 mg: Blinded Phase: Participants received SIM 200 mg administered via intravenous infusion every 2 weeks for up to 240 weeks.
  Open-Label Phase: Participants received SIM 700 mg administered via intravenous infusion every 2 weeks for up to an additional 240 weeks.
- Total: Total of all reporting groups
Arm/Group | SIM 200 mg | SIM 700 mg | Placebo | Total
Number analyzed (Participants) | 87 | 86 | 85 | 258
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (7.2) | 55 (7.3) | 56 (7.8) | 55 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 54 | 56 | 163
  Male | 34 | 32 | 29 | 95
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 3 | 1 | 0 | 4
  Race: Black | 2 | 3 | 1 | 6
  Race: White | 80 | 75 | 83 | 238
  Race: Other | 2 | 7 | 1 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 12 | 17 | 10 | 39
  Ethnicity: Not Hispanic or Latino | 75 | 69 | 75 | 219
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 67 | 68 | 76 | 211
  France | 6 | 4 | 3 | 13
  Canada | 5 | 1 | 2 | 8
  Germany | 1 | 4 | 3 | 8
  Spain | 3 | 5 | 0 | 8
  United Kingdom | 3 | 3 | 1 | 7
  Italy | 2 | 1 | 0 | 3
Hepatic Venous Pressure Gradient (HVPG) [Mean (Standard Deviation); unit: mmHg] — Population: Full Analysis Set included all enrolled participants who were randomized and received at least 1 dose of study drug. Only participants with available baseline data were analyzed.
  mmHg
    number analyzed (Participants) | 87 | 85 | 84 | 256
    (all) | 12.9 (5.10) | 12.8 (5.37) | 13.0 (5.25) | 12.9 (5.22)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hepatic Venous Pressure Gradient (HVPG)
Time Frame: Baseline to Week 96
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | SIM 200 mg | SIM 700 mg | Placebo
Number analyzed (Participants) | 63 | 66 | 68
mmHg | -0.1 (3.76) | 0.0 (4.23) | -0.1 (4.01)
Statistical Analysis 1: Comparison: SIM 200 mg vs Placebo; A mixed-effect model for repeated measures (MMRM) with an unstructured variance-covariance matrix for each participant was used to calculate a point estimate and a 95% confidence interval (CI) for the treatment difference between each treatment arm and placebo in least squares mean (LSMean) change from baseline in HVPG at Week 96. With MMRM setting, all participants with available data from 3 treatment groups with change in HVPG at Week 96 contributed to the overall model; Test type: Superiority; Difference in LSMeans [SIM - Placebo] = 0.1, 95% CI 2-sided [-1.2 to 1.5]
Statistical Analysis 2: Comparison: SIM 700 mg vs Placebo; An MMRM with an unstructured variance-covariance matrix for each participant was used to calculate a point estimate and a 95% CI for the treatment difference between each treatment arm and placebo in LSMean change from baseline in HVPG at Week 96. With MMRM setting, all participants with available data from 3 treatment groups with change in HVPG at Week 96 contributed to the overall model; Test type: Superiority; Difference in LSMeans [SIM - Placebo] = 0.1, 95% CI 2-sided [-1.2 to 1.4]

2. Primary Outcome: Event-Free Survival (EFS) Using Kaplan-Meier
Description: Event free survival (EFS) was the primary clinical efficacy endpoint and was assessed by time to first liver-related event or death, whichever occurs first. Liver-related events included any of the following:
  * Liver transplantation
  * Qualification for liver transplantation
  * Model for End-Stage Liver Disease (MELD) ≥ 15
  * Events indicative of hepatic decompensation
  * Esophageal variceal bleeding
  * Ascites
  * Hepatic Encephalopathy
  * ≥ 2 point increase in Child Pugh-Turcotte (CPT) score
  * Newly diagnosed varices in a subject without prior varices
Time Frame: Baseline up to the time of clinical event or last dose date (maximum: 240 weeks in Blinded Phase); which ever occurred first
Population: Participants in the Full Analysis Set were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | SIM 200 mg | SIM 700 mg | Placebo
Number analyzed (Participants) | 87 | 86 | 85
months | NA [NA to NA] — Data was not estimable as more than 50% of participants were censored. | NA [NA to NA] — Data was not estimable as more than 50% of participants were censored. | NA [NA to NA] — Data was not estimable as more than 50% of participants were censored.
Statistical Analysis 1: Comparison: SIM 200 mg vs Placebo; Differences in EFS between a given SIM group and placebo were assessed using the log-rank test stratified by HVPG category (< 10 mmHg vs ≥ 10 mmHg) and presence or absence of diabetes at baseline; Test type: Superiority; p = 0.41, Stratified log-rank test
Statistical Analysis 2: Comparison: SIM 700 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.065, Stratified log-rank test

ADVERSE EVENTS:
Time Frame: Baseline up to the last dose date plus 30 days (average exposure: SIM 200 mg= 109.3 weeks, SIM 700 mg= 115.9 weeks, Placebo= 120.2 weeks, Open-label SIM 700 mg= 46.2 weeks)
Description: Safety Analysis Set included all enrolled participants who were randomized and received at least one dose of study drug and Open-Label Safety Analysis Set included all participants who rolled over into the open-label phase and received at least 1 dose of open-label study drug.
Groups:
- Blinded Phase: SIM 200 mg: Adverse events recorded in this group occurred during the Blinded Phase. Participants received SIM 200 mg administered via intravenous infusion every 2 weeks for up to 240 weeks.
- Blinded Phase: SIM 700 mg: Adverse events recorded in this group occurred during the Blinded Phase. Participants received SIM 700 mg administered via intravenous infusion every 2 weeks for up to 240 weeks.
- Blinded Phase: Placebo: Adverse events recorded in this group occurred during the Blinded Phase. Participants received placebo to match SIM administered via intravenous infusion every 2 weeks for up to 240 weeks.
- Open-Label Phase: SIM 700 mg: All participants who completed the randomized phase through the Week 240 visit, or who had an adjudicated clinical event prior to completing the randomized phase, were offered the opportunity to receive open-label SIM for up to 240 additional weeks. Adverse events recorded in this group occurred during the Open-Label Phase. All participants received fixed-dose open-label SIM 700 mg intravenous infusions every 2 weeks for up to 240 weeks.
Arm/Group | Blinded Phase: SIM 200 mg | Blinded Phase: SIM 700 mg | Blinded Phase: Placebo | Open-Label Phase: SIM 700 mg
Serious Adverse Events (participants affected / at risk) | 37/87 | 36/86 | 25/85 | 17/40
Other Adverse Events (participants affected / at risk) | 85/87 | 81/86 | 83/85 | 32/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Blinded Phase: SIM 200 mg (N=87) | Blinded Phase: SIM 700 mg (N=86) | Blinded Phase: Placebo (N=85) | Open-Label Phase: SIM 700 mg (N=40)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Bandaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 1 | 0 | 0
Atrioventricular block second degree (Cardiac disorders) | 1 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 0 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 1 | 1 | 0 | 0
Basedow's disease (Endocrine disorders) | 0 | 1 | 0 | 0
Hyperparathyroidism (Endocrine disorders) | 0 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 2 | 3 | 1 | 2
Colitis (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diverticulum (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Epiploic appendagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 2 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Hernial eventration (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 | 2 | 2 | 1
Pancreatitis (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Varices oesophageal (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 1
Chest pain (General disorders) | 3 | 2 | 2 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0
Peripheral swelling (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0
Systemic inflammatory response syndrome (General disorders) | 0 | 1 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Gallbladder polyp (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Haemobilia (Hepatobiliary disorders) | 0 | 1 | 1 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Ischaemic hepatitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0
Bacterial pyelonephritis (Infections and infestations) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 2 | 1 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 1 | 1
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0
Escherichia sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis bacterial (Infections and infestations) | 0 | 0 | 0 | 1
Kidney infection (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 2 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1 | 0
Rocky mountain spotted fever (Infections and infestations) | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 3 | 2 | 0
Urinary tract infection (Infections and infestations) | 3 | 1 | 2 | 0
Viral infection (Infections and infestations) | 1 | 1 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Post procedural discomfort (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Procedural hypotension (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Blood osmolarity decreased (Investigations) | 0 | 0 | 0 | 1
Electrocardiogram T wave peaked (Investigations) | 0 | 0 | 0 | 1
Model for end stage liver disease score abnormal (Investigations) | 0 | 0 | 0 | 1
Model for end stage liver disease score increased (Investigations) | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 2
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 2
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Altered state of consciousness (Nervous system disorders) | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 1
Cervical myelopathy (Nervous system disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 3 | 4 | 2 | 5
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0
Migraine with aura (Nervous system disorders) | 1 | 0 | 0 | 0
Nerve compression (Nervous system disorders) | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 2 | 0
Temporal lobe epilepsy (Nervous system disorders) | 1 | 0 | 0 | 0
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Drug abuse (Psychiatric disorders) | 0 | 0 | 1 | 0
Major depression (Psychiatric disorders) | 0 | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 1 | 0 | 0 | 0
Psychiatric decompensation (Psychiatric disorders) | 0 | 0 | 0 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 1 | 2 | 3
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0 | 0
Ureterolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
Hepatic hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 1
Portopulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 2 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Blinded Phase: SIM 200 mg (N=87) | Blinded Phase: SIM 700 mg (N=86) | Blinded Phase: Placebo (N=85) | Open-Label Phase: SIM 700 mg (N=40)
Anaemia (Blood and lymphatic system disorders) | 10 | 7 | 6 | 3
Splenomegaly (Blood and lymphatic system disorders) | 3 | 4 | 6 | 0
Palpitations (Cardiac disorders) | 6 | 1 | 3 | 0
Vertigo (Ear and labyrinth disorders) | 4 | 6 | 5 | 0
Abdominal distension (Gastrointestinal disorders) | 9 | 10 | 9 | 4
Abdominal pain (Gastrointestinal disorders) | 19 | 23 | 14 | 5
Abdominal pain lower (Gastrointestinal disorders) | 5 | 3 | 4 | 0
Abdominal pain upper (Gastrointestinal disorders) | 15 | 19 | 13 | 5
Ascites (Gastrointestinal disorders) | 7 | 8 | 9 | 7
Constipation (Gastrointestinal disorders) | 9 | 15 | 10 | 2
Diarrhoea (Gastrointestinal disorders) | 24 | 23 | 33 | 7
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 | 4 | 3 | 1
Haemorrhoids (Gastrointestinal disorders) | 3 | 2 | 5 | 1
Nausea (Gastrointestinal disorders) | 29 | 28 | 28 | 9
Portal hypertensive gastropathy (Gastrointestinal disorders) | 1 | 0 | 8 | 1
Umbilical hernia (Gastrointestinal disorders) | 1 | 1 | 0 | 2
Varices oesophageal (Gastrointestinal disorders) | 5 | 10 | 8 | 0
Vomiting (Gastrointestinal disorders) | 13 | 15 | 19 | 6
Asthenia (General disorders) | 3 | 5 | 5 | 3
Chest pain (General disorders) | 8 | 10 | 6 | 1
Chills (General disorders) | 3 | 5 | 4 | 1
Fatigue (General disorders) | 34 | 32 | 28 | 6
Infusion site pain (General disorders) | 7 | 0 | 6 | 0
Oedema peripheral (General disorders) | 13 | 14 | 16 | 6
Pain (General disorders) | 7 | 6 | 3 | 1
Peripheral swelling (General disorders) | 8 | 7 | 6 | 2
Pyrexia (General disorders) | 10 | 9 | 6 | 3
Cholelithiasis (Hepatobiliary disorders) | 1 | 2 | 7 | 0
Hepatomegaly (Hepatobiliary disorders) | 3 | 2 | 7 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 2
Bronchitis (Infections and infestations) | 14 | 14 | 15 | 2
Gastroenteritis (Infections and infestations) | 6 | 4 | 2 | 1
Gastroenteritis viral (Infections and infestations) | 5 | 1 | 2 | 1
Herpes zoster (Infections and infestations) | 5 | 2 | 1 | 1
Influenza (Infections and infestations) | 4 | 6 | 8 | 2
Localised infection (Infections and infestations) | 1 | 1 | 2 | 2
Nasopharyngitis (Infections and infestations) | 15 | 16 | 19 | 2
Peritonitis bacterial (Infections and infestations) | 0 | 0 | 0 | 2
Pneumonia (Infections and infestations) | 2 | 5 | 2 | 2
Sinusitis (Infections and infestations) | 14 | 16 | 17 | 3
Upper respiratory tract infection (Infections and infestations) | 15 | 19 | 11 | 3
Urinary tract infection (Infections and infestations) | 9 | 14 | 18 | 3
Contusion (Injury, poisoning and procedural complications) | 10 | 6 | 16 | 5
Fall (Injury, poisoning and procedural complications) | 7 | 5 | 13 | 4
Infusion related reaction (Injury, poisoning and procedural complications) | 10 | 7 | 11 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 5 | 4 | 2 | 0
Muscle strain (Injury, poisoning and procedural complications) | 5 | 1 | 4 | 0
Procedural pain (Injury, poisoning and procedural complications) | 8 | 7 | 7 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 2
Skin abrasion (Injury, poisoning and procedural complications) | 4 | 1 | 2 | 2
Blood creatinine increased (Investigations) | 1 | 1 | 5 | 0
Blood glucose increased (Investigations) | 2 | 1 | 5 | 2
Weight increased (Investigations) | 4 | 1 | 5 | 0
Decreased appetite (Metabolism and nutrition disorders) | 7 | 2 | 11 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 10 | 6 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 2 | 2 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 3 | 2 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1 | 2 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 | 19 | 13 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 27 | 18 | 12 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 3 | 5 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 7 | 4 | 2 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 16 | 13 | 10 | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 10 | 6 | 7 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 2 | 8 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 8 | 3 | 5 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 | 9 | 9 | 1
Dizziness (Nervous system disorders) | 14 | 8 | 9 | 2
Headache (Nervous system disorders) | 26 | 28 | 17 | 5
Hepatic encephalopathy (Nervous system disorders) | 7 | 6 | 6 | 4
Syncope (Nervous system disorders) | 4 | 1 | 2 | 2
Tremor (Nervous system disorders) | 4 | 4 | 5 | 0
Anxiety (Psychiatric disorders) | 7 | 3 | 3 | 1
Depression (Psychiatric disorders) | 4 | 7 | 2 | 2
Insomnia (Psychiatric disorders) | 7 | 5 | 9 | 2
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 1 | 2
Dysuria (Renal and urinary disorders) | 1 | 1 | 3 | 3
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 2 | 2
Gynaecomastia (Reproductive system and breast disorders) | 2 | 0 | 1 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 16 | 12 | 13 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 6 | 4 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 | 9 | 6 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 7 | 7 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 11 | 8 | 9 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 7 | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 6 | 3 | 3 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 9 | 11 | 6 | 3
Rash (Skin and subcutaneous tissue disorders) | 8 | 11 | 15 | 0
Hypertension (Vascular disorders) | 6 | 3 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years